CLINICAL TRIAL: NCT00348465
Title: An Observational Study to Evaluate the Changes in Prostate Volume Over Time With The Use of Transrectal Ultrasound and Computed Tomography Following Permanent Prostate Brachytherapy With Iodine-125 Seeds.
Brief Title: Prostate Volume Changes Following Prostate Brachytherapy With Iodine-125 Seeds
Status: Completed | Type: Observational
Sponsor: New York Presbyterian Brooklyn Methodist Hospital (Other)
Responsible Party: Principal Investigator, Hani Ashamalla, MD, MD, New York Presbyterian Brooklyn Methodist Hospital
Other Study IDs: NYM-353
Record Dates: First submitted 2006-07-03; First posted 2006-07-04 (Estimated); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Prostate Cancer
Keywords: Brachytherapy; Prostate volume
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Brachytherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Brachytherapy with Iodine-125 seeds — Brachytherapy of the prostate, and measurements of the prostate volume using CT scan and TURS
  Other Names: Prostate Volume over time

SUMMARY:
The size of the prostate changes due to insertion of the radioactive seeds. We will measure the prostate size, before and after the procedure.

DETAILED DESCRIPTION:
The prostate size will be measured using the TRUS and CT scan on days -1, 0, 1, 9, 30, and 60 days after the brachytherapy procedure.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of prostate cancer
* T1-3 disease
* PSA <20 ng/ml
* Patient must sign a study-specific informed consent prior to enrollment.

Exclusion Criteria:

* Patients ineligible to brachytherapy

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prostate Cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2006-05 (Actual); Primary Completion 2007-12 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hani Ashamalla, MD, FCCP, Study Chair — New York Presbyterian Brooklyn Methodist Hospital; Ewa Bieniek, MD, Principal Investigator — NY Methodist Hospital